CLINICAL TRIAL: NCT05591872
Title: Low Dose Versus High Dose Heparin With or Without Hemostasis Patch and Radial Access Site Outcomes; an Open-label Factorial Randomized Trial (InnoSEAL III)
Brief Title: Low Dose Heparin Factorial Trial
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tabba Heart Institute (Other)
Collaborators: InnoTherapy Inc (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: THI-INNOSEAL3-2022
Record Dates: First submitted 2022-10-19; First posted 2022-10-24 (Actual); Last update posted 2022-10-24 (Actual); Status verified 2022-10

CONDITIONS: Radial Artery Occlusion
Keywords: radial artery occlusion, left heart catheterization, heparin, hemostatic patch
MeSH Terms: conditions — Arterial Occlusive Diseases

STUDY DESIGN:
Intervention Model Description: 2x2 Heparin: Low dose (LD) vs. standard dose (SD) Device type: InnoSEAL + TRBand (I+TRB) vs. TRBand alone (TRB)
  Intervention arms:
  1. LD+I+TRB
  2. LD+TRB
  3. SD+I+TRB
  4. SD+TRB
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- LD+I+TRB (Active Comparator): Patient will get heparin dose according to their weight i.e. (<60 Kg-2000 IU; 60-80 Kg-2500 IU; >80 Kg-3000 IU)
  And access site will be secured with InnoSEAL patch plus TRB
  Interventions: Drug: LD+I+TRB
- LD+TRB (Active Comparator): Patient will get heparin dose according to their weight i.e. (<60 Kg-2000 IU; 60-80 Kg-2500 IU; >80 Kg-3000 IU)
  And access site will be secured with TRB alone
  Interventions: Drug: LD+I+TRB
- SD+I+TRB (Active Comparator): Patient will get standard heparin dose of 5000 IU.
  And access site will be secured with InnoSEAL patch plus TRB
  Interventions: Drug: LD+I+TRB
- SD+TRB (No Intervention): This is the control arm. Patient will get standard heparin dose of 5000 IU.
  And access site will be secured with TRB.

INTERVENTIONS:
Drug: LD+I+TRB — Same as in the arm description
  Other Names: SD+I+TRB; LD+TRB
  Arms: LD+I+TRB; LD+TRB; SD+I+TRB

SUMMARY:
An open label 2x2 factorial randomized trial is planned to determine the difference in mean hemostasis time between low dose heparin (LD) i.e between 2000-3000 IU and standard dose heparin (SD) i.e. 5000 IU with or without catecholamine chitosan-based pad (InnoSEAL hemostatic pad, InnoTherapy, Inc. S Korea) used in conjunction with TRB (InnoSEAL+TRB [I+TRB]) among patients who are undergoing left heart cath at Tabba Heart Institute.

Secondary objectives include testing the difference in radial artery occlusion (RAO), and hematoma (III, IV grade) and composite outcome (RAO+hematoma).

DETAILED DESCRIPTION:
Eligibility criteria:

Hemodynamically stable adult patients of both genders, who will undergo transradial coronary angiogram (CAG) using 6 F sheath will be included. Patients who had STEMI, are on anticoagulants after procedure or on an ongoing anticoagulation therapy, have ipsilateral arteriovenous fistula, RAO at baseline, Barbeau's class D will be excluded.

Intervention:

After written consent, first randomization will be done to the heparin arm. If participant falls in LD heparin group, he/she will receive IV heparin 2000-3000 IU (<60 Kg-2000 IU; 60-80 Kg-2500 IU; >80 Kg-3000 IU) at the start of CAG and if SD then 5000 IU of heparin will be administered. Second randomization will be done to allocate the participant in I+TRB or TRB alone arm.

In I+TRB arm, after the completion of CAG, at radial artery site, the sheath is pulled 2-3cm and the area surrounding the puncture site is cleaned, dried and InnoSEAL is placed over the puncture site. A transparent adhesive clear dressing is placed over the InnoSEAL and TRB is applied over the dressing.

In TRB arm, TRB alone will be applied over the puncture site. In both the arms, 10 cc air will be inserted in TRB at the start of the protocol, then at 10, 20, and 30 minutes after the procedure 2cc, then 4cc, and then 6cc or remaining air will be withdrawn. If patient oozes or bleeds from radial site in between the protocol, 2 cc air or more will be inserted to control the bleeding. After reaching 0cc air in TRB, deflated TRB will be observed for 15 minutes. The TRB will be removed and access site will further be observed for 15 minutes for hematoma, oozing/bleeding.

At each air draw, reverse Barbeau's test will be done to check the radial artery occlusion. If radial pulse is found absent after removing TRB, then radial artery colored doppler ultrasound will be done to confirm the radial artery occlusion.

The time from the removal of radial sheath till removal of TRB will be recorded as the compression time needed to achieve hemostasis at the radial access site.

ELIGIBILITY:
Inclusion Criteria:

* Hemodynamically stable adult patients of both genders, who will undergo transradial coronary angiogram (CAG) using 6 F sheath will be included.

Exclusion Criteria:

* Patients who had STEMI, are on anticoagulants after procedure or on an ongoing anticoagulation therapy, have ipsilateral arteriovenous fistula, RAO at baseline, Barbeau's class D will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2022-05-09 (Actual); Primary Completion 2023-04-30 (Estimated); Study Completion 2023-10-31 (Estimated)

PRIMARY OUTCOMES:
Compression time | 45 minutes
  Time from radial sheath removal to the time of TRB removal

SECONDARY OUTCOMES:
radial artery occlusion | 24 hours
  Radial artery occlusion on colored doppler ultrasound
Hematoma at the access site | 24 hours
  Hematoma will be graded according to BRAC and BRAC III or IV will be considered as significant hematoma.

CONTACTS AND LOCATIONS:
Overall Officials: Sana Sheikh, M.Sc, Study Director — Tabba Heart Institute
Locations (1):
- Sana, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No
Individual data will not be shared.